CLINICAL TRIAL: NCT02543216
Title: Gene - Diet Interactions in Fatty Acid Desaturase 1 Gene (FADSDIET)
Brief Title: Gene - Diet Interactions in Fatty Acid Desaturase 1 Gene
Acronym: FADSDIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Jussi Pihlajamäki, Professor, University of Eastern Finland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FADSDIET
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Fatty Acid
Keywords: fatty acids, FADS gene, genotype, diet
MeSH Terms: interventions — Sunflower Oil

ARMS (2):
- CC genotype (Experimental): 4-week study diets were isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (25-45 g) sunflower oil daily depending on body weight. The same diets were instructed for both genotypes.
  Interventions: Dietary Supplement: Sunflower oil
- TT genotype (Experimental): 4-week study diets were isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (25-45 g) sunflower oil daily depending on body weight. The same diets were instructed for both genotypes.
  Interventions: Dietary Supplement: Sunflower oil

INTERVENTIONS:
Dietary Supplement: Sunflower oil — Study diets were isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (25-45 g) sunflower oil daily depending on body weight. Thus, approximately 16-28 g (6 E%) LA were provided daily on top of the average intake of approximately 10-12 g (4.5 E%).

SUMMARY:
Interactions between genes and environment, are likely to be crucial in the development of the common diseases such as type 2 diabetes. It was recently shown that FADS1 and FADS 2 genotypes are the strongest genes in a genome-wide analysis regulating serum fatty acid profile.The aim of this study is to test if subjects with the CC and TT genotypes of the FADS1 gene (rs174547) respond differentially to a diet supplemented with linoleic acid (substrate for FADS). We hypothesize that subjects with the TT genotype with more active desaturases will be more sensitive to dietary modification leading to more robust differences in serum FA profile, tissue inflammation and serum lipids.

DETAILED DESCRIPTION:
Lean and overweight subjects (BMI >20kg/m2 <29kg/m2 ) with CC and TT genotypes of FADS1 polymorphism (rs174547) were recruited from the METSIM study (METabolic Syndrome in Men, currently >10000 men included from the population living in Kuopio). The potential participants were asked to contact study nurse if willing to participate. Twenty six subjects with CC genotype were selected after matching with thirty six subjects with the TT genotype for age, BMI and medication.

Study diet were isocaloric following the habitual diet of the participants with a supplement of 30-50 ml (25-45 g) sunflower oil daily depending on body weight. Thus, approximately 16-28 g (6 E%) LA daily were provided on top of the average intake of approximately 10-12 g (4.5 E%). This dose of sunflower oil is not known to cause any side effects or adverse events and even higher doses have been safe.

Food records were collected at the beginning (4 days) and during the third week of the study (7 days) to estimate daily intake of macronutrients and specifically of different fatty acids.

ELIGIBILITY:
Inclusion Criteria:

Participant of Metabolic syndrome in men (METSIM) cohort BMI 20-30 kg/m2 Healthy CC/TT genotype (rs 174547)

Exclusion Criteria:

Type 2 diabetes Other chronic disease

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Fatty acid profile of serum lipid fractions | 4 weeks

SECONDARY OUTCOMES:
Serum lipids an lipoproteins | 4 weeks
Adipose tissue biopsies | 4 weeks
white blood cell samples | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Eastern Finland, Clinical Nutrition, Kuopio, Finland

REFERENCES:
- [Derived] Meuronen T, Lankinen MA, Karkkainen O, Laakso M, Pihlajamaki J, Hanhineva K, Schwab U. FADS1 rs174550 genotype and high linoleic acid diet modify plasma PUFA phospholipids in a dietary intervention study. Eur J Nutr. 2022 Mar;61(2):1109-1120. doi: 10.1007/s00394-021-02722-w. Epub 2021 Oct 31. PMID 34718859
- [Derived] Lankinen MA, Fauland A, Shimizu BI, Agren J, Wheelock CE, Laakso M, Schwab U, Pihlajamaki J. Inflammatory response to dietary linoleic acid depends on FADS1 genotype. Am J Clin Nutr. 2019 Jan 1;109(1):165-175. doi: 10.1093/ajcn/nqy287. PMID 30624587